CLINICAL TRIAL: NCT05823961
Title: Interventional, Non-comparative, Single-center PMCF Study to Evaluate Performance and Safety of "Cross-Linked Hyaluronic Acid (CLHA)-Based Eyedrops" Used to Improve Lacrimal Abnormalities, Even When Associated With Dry Eye Symptoms
Brief Title: PMCF Study to Evaluate Performance and Safety of "CLHA-based Eyedrops" Used to Improve Lacrimal Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.O.C. Farmaceutici S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COC-R5-CLHA
Record Dates: First submitted 2023-04-11; First posted 2023-04-21 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-05

CONDITIONS: Dry Eye Disease; Dry Eye; Kerato Conjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyedrops treatment arm (Experimental)
  Interventions: Device: Cross-linked hyaluronic acid eye drops

INTERVENTIONS:
Device: Cross-linked hyaluronic acid eye drops — Cross-linked hyaluronic acid (CLHA)-based eyedrops

SUMMARY:
Tear dysfunction, also known as Dry Eye Disease (DED) is frequently encountered in the clinical practice. It is a multifactorial disease of the ocular surface characterized by insufficient tear production, loss of homeostasis of the tear film, increased osmotic stress of the ocular surface, ocular discomfort and visual disturbance.

Hyaluronic acid (HA) is a linear heteropolysaccharide (glycosaminoglycan) with unique hygroscopic, rheological, and lubricating properties. HA is naturally found at the human ocular surface where it contributes to the ocular hydration and lubrication thanks to its capability to bind water molecules.Sodium hyaluronate (SH), the salt form of HA, is widely used in artificial tears to counteract dry eye symptoms by facilitating eyelid sliding and reducing its friction on the corneal-conjunctival surface.

Conventional HA-based eye drops contain linear HA. However, artificially cross-linked HA (CLHA) has several advantages over linear HA in alleviating dry eye symptoms. The increased viscoelasticity of CLHA results in a greater stability and a better resistance to the enzymatic degradation by hyaluronidase, while preserving all the properties of linear HA. Furthermore, chemical cross-linking of HA extends its permanence on the ocular surface, thus reducing the number of instillations and increasing patients' compliance.

For these reasons, an interventional, non-comparative, single-center Post Marketing Clinical Follow-up (PMCF) study was planned to evaluate the performance and safety of "Cross-Linked Hyaluronic Acid (CLHA)-based eyedrops" used as intended to improve lacrimal abnormalities, even when associated with dry eye symptoms.

The objectives of the PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with use of "Cross-Linked Hyaluronic Acid (CLHA)-based eyedrops" according to the Instructions for Use (IFU).

Each subject, after signing the Informed Consent Form (ICF), will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit (V0), one of the "CLHA-based eyedrops" products will be administered to the enrolled subject.

The patient will perform 2 on-site visits: V0 and V2/EOS. To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events and concomitant medications intake.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed;
* Male and Female Aged ≥ 18 years at the time of the signature of the ICF;
* Patients with dry eye symptoms and/or redness, fatigue, discomfort of the eye or the ocular mucosa due to intrinsic or extrinsic factors such as atmospheric agents, environmental factors, inflammation, blepharitis, eye surgery, and/or use of contact lenses;
* Willing not to use other eye drops during the entire treatment period.

Exclusion Criteria:

* Other - different - eyes clinical conditions (e.g. glaucoma);
* Suspected alcohol or drug abuse;
* Known hypersensitivity or allergy to Investigational Product (IP) components;
* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. rheumatic diseases, diabetes);
* Participation in another investigational study;
* Inability to follow all study procedures, including attending all site visits, tests and examinations;
* Mental incapacity that precludes adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Change in Schirmer Test I: to evaluate the performance of the "CLHA-based eyedrops" used to improve lacrimal abnormalities, even when associated with dry eye symptoms due to intrinsic or extrinsic factors, through the Schirmer I test | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI): to evaluate the performance of the "CLHA-based eyedrops" used to relieve discomfort to the eyes or ocular mucosa, and eye fatigue caused by intrinsic or extrinsic factors, through OSDI | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)
Change in Tear Break-up Time (TBUT): to evaluate the performance of the "CLHA-based eyedrops" used to improve tear film stability in subjects with dry eye symptoms and/or after eye surgery, through the TBUT test | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)
The global patient treatment tolerance to the "Cross-Linked Hyaluronic Acid (CLHA)-based eyedrops" as assessed by the Visual Analogue Scale (VAS) as a difference between baseline and Day 30. | End of study visit (EOS/V2 = Day 30 ± 2)
  Visual Analogue Scale:
  Minimum value = 0; Maximum value = 10; Higher scores mean a better outcome.
To evaluate the patient satisfaction through a Rensis Likert 5 points patient satisfaction scale | End of study visit (EOS/V2 = Day 30 ± 2)
  Rensis Likert 5 points patient satisfaction scale Minimum value: Very dissatisfied Maximum value: Very satisfied Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria Policlinico "G.Rodolico - San Marco", Catania, CT, Italy